CLINICAL TRIAL: NCT05788263
Title: The Effects of Neuroscience-Based Exercise Approaches on Pain, Disability and Gait Parameters in Individuals With Chronic Non-Specific Neck Pain
Brief Title: The Effects of Neuroscience-Based Exercise
Acronym: NBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Tekin (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Sponsor-Investigator, Fatih Tekin, Assist. Prof., Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEUROSCİENCE
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Chronic Neck Pain; Persistent Neck Pain; Neuroscience Approach
Keywords: Neuroscience based exercises; Chronic neck pain; gait parameters

STUDY DESIGN:
Intervention Model Description: basic randomization via spss 24.00 program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Craniovertebral angle assesment (Experimental): Craniovertebral angle is the most widely used measurement to assess Forward head posture. Craniovertebral angle is described as the acute angle formed between a horizontal line passing through the spinous process of the seventh cervical vertebra (C7) and the line connecting the midpoint of the tragus to the spinous process of C7.
  Interventions: Other: neuroscience based aproach
- Spatio-temporal gait analyz (LEGSystm) (Experimental): The gait performance of the cases was evaluated with a spatio-temporal gait analysis device named LEGSystm developed by BioSensicstm. The device consists of two sensors. The sensors are placed 3-5 cm above the ankle of the subject to be tested with the help of velcro. The device is controlled from the computer with its own software and instantly sends the raw data it collects to the computer via Bluetooth. The software analyzes the raw data it receives from the device and turns it into results.The Modified Get Up and Go Test (MKYT), which is also supported by the legsyst, was used for assesment. The test was repeated 2 times and the average time was recorded. Legsystm provides information on double stride length, duration and speed of walking, as well as standing, turning, sitting times and total time
  Interventions: Other: neuroscience based aproach
- Neck Disabilty Index (Experimental): It is a questionnaire created to determine the level of disability caused by chronic neck pain in daily life.
  Interventions: Other: neuroscience based aproach

INTERVENTIONS:
Other: neuroscience based aproach — exercise for pain

SUMMARY:
The aim of this study is to examine the effects of neuroscience-based exercise approaches on pain, disability and gait parameters in individuals with non-specific chronic neck pain.

Material- Methods Demographic data, gait parameters, Dizabilty level and craniovertebral angle values of individuals were evaluated with clinical data evaluation form, Spatio-Temporal Gait Analysis (LEGSystm), Neck Disability Index and photometer, respectively. The evaluations were performed 2 times before and after the treatment.

DETAILED DESCRIPTION:
Neuroscience-based exercise approaches are a promising method that has been introduced in recent years in the treatment of non-specific musculoskeletal pain and related dysfunctions. The basis of this method is the exercises and trainings created by considering the neurobiological (changes in tissues) and neurophysiological basis (brain fog, somatosensory sensitization) of nociplastic pain in the musculoskeletal system. In the neuroscience-based exercise approach, it is aimed to reduce the increase in sensitivity in brain fog and somatosensory pathways. The main purpose is to teach the cortex that movement can be done painlessly and accurately and to alleviate the symptoms in the related tissues. It is aimed to perform the exercise painlessly and accurately by adding cognitive goals and changing the focus (14). In the literature, although there are very few studies showing that neuroscience education and therapeutic exercise combinations are effective on chronic nociplastic pain in patients with non-specific chronic neck pain, no studies examining the effects of neuroscience-based exercise approaches on gait parameters in individuals with non-specific chronic neck pain were found (15). ,16). Our study will contribute to the literature in this field and will reveal the effects of neuroscience-based exercise approaches more clearly. The aim of this study is to examine the effects of neuroscience-based exercise approaches on pain, disability and gait parameters in individuals with non-specific chronic neck pain.

Material- Methods Demographic data, gait parameters, Dizabilty level and craniovertebral angle values of individuals were evaluated with clinical data evaluation form, Spatio-Temporal Gait Analysis (LEGSystm), Neck Disability Index and photometer, respectively. The evaluations were performed 2 times before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing with chronic non-specific neck pain
* Volunteer to participate in the study
* beetwen 18-25 years old

Exclusion Criteria:

* have had any cervical area surgery
* having any disease that would affect the assessments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
craniovertebral angle degree | 1 minute
  Craniovertebral angle is the most widely used measurement to assess Forward head posture. Craniovertebral angle is described as the acute angle formed between a horizontal line passing through the spinous process of the seventh cervical vertebra (C7) and the line connecting the midpoint of the tragus to the spinous process of C7.
Legsystm | 1 minute
  The gait performance of the cases was evaluated with a spatio-temporal gait analysis device named LEGSystm developed by BioSensicstm. The device consists of two sensors. The sensors are placed 3-5 cm above the ankle of the subject to be tested with the help of velcro. The device is controlled from the computer with its own software and instantly sends the raw data it collects to the computer via Bluetooth. The software analyzes the raw data it receives from the device and turns it into results.The Modified Get Up and Go Test (MKYT), which is also supported by the legsyst, was used for assesment. The test was repeated 2 times and the average time was recorded. Legsystm provides information on double stride length, duration and speed of walking, as well as standing, turning, sitting times and total time.
Neck Disability Index | 3 minutes
  It is a questionnaire created to determine the level of disability caused by chronic neck pain in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: fatih tekin, assist prof, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No